CLINICAL TRIAL: NCT03326102
Title: A Multi-national,Multi-center, Open-label, Phase 2 Clinical Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of DHP107 (Liporaxel®,Oral Paclitaxel) Compared to IV Paclitaxel in Patients With Recurrent or Metastatic Breast Cancer(OPERA)
Brief Title: Oral Paclitaxel Efficacy Safety and PK in Recurrent and Metastatic Breast Cancer
Acronym: OPERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107CS-6
Record Dates: First submitted 2017-10-19; First posted 2017-10-30 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2022-01

CONDITIONS: Recurrent or Metastatic Breast Cancer
Keywords: Breast Cancer; DHP107; Paclitaxel; Liporaxel
MeSH Terms: conditions — Recurrence; Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to DHP107 or IV paclitaxel in a ratio of 2:1 (n=48 to DHP107 and n=24 to IV paclitaxel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DHP107 (Experimental): The 12 eligible subjects will receive DHP107 and be taken blood samples for PK analysis on Day 1, 8 of cycle 1.
  Total 48 subjects (including PK subjects) will receive DHP107 200 mg/m2 orally twice daily on Days 1, 8 and 15 every 28 days.
  Interventions: Drug: DHP107
- IV paclitaxel (Experimental): Total 24 subject will receive IV paclitaxel 80 mg/m2 weekly.(3 weeks on/1 week off)
  Interventions: Drug: IV Paclitaxel

INTERVENTIONS:
Drug: DHP107 — DHP107 200mg/m2 orally twice daily on Days 1, 8 and 15 every 28 days
  Other Names: Liporaxel®, Oral Paclitaxel
  Arms: DHP107
Drug: IV Paclitaxel — IV Paclitaxel 80 mg/m2 QW (3 weeks on/1 week off)
  Other Names: Taxol Injection
  Arms: IV paclitaxel

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and pharmacokinetics of DHP107 (Oral Paclitaxel, Korea brand name: Liporaxel®) compared to IV Paclitaxel in patients with Recurrent or Metastatic Breast Cancer.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with confirmed diagnosis of recurrent or metastatic breast cancer based on histopathology examination
2. Subjects with diagnosis of HER2-negative breast cancer that was confirmed by IHC or in situ hybridization (ISH) assessment of tumor samples
3. Subjects who have received up to 3 lines of therapy for advanced disease, without prior exposure to taxane in the advanced stage setting
4. Subjects who have a performance status of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale.
5. Subjects who have measurable disease according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST version 1.1).

Key Exclusion Criteria:

1. Subjects who have received prior taxane therapy in the metastatic setting
2. Subjects whose adjuvant or neoadjuvant treatment for early stage breast cancer was completed within 6 months prior to entry into the study.
3. Subjects with neuropathy grade ≥2 based on CTCAE v4.03 at the time of study entry
4. Subjects with symptomatic, untreated metastases to the central nervous system (CNS) at the time of screening.
5. Subjects who have received any investigational drugs or devices within 4 weeks before the first day of study treatment (C1D1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Every 8 weeks upto 18 months from randomization date
  ORR is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1) criteria

SECONDARY OUTCOMES:
Progression free survival(PFS) | Up to 18 months from randomization date
  PFS is defined as the time from date of randomization until the date of first documented progression or death.
Overall survival(OS) | Up to 36 months from FPI
  OS is defined as the time from the date of inclusion to the date of death.
Time to treatment failure(TTF) | Up to 18 months from randomization date
  TTF is defined as the time from the randomization date to the date of discontinuation of treatment, regardless of the cause.
Duration of response(DOR) | Up to 18 months from randomization date
  DOR is the time between the initial response to therapy and subsequent disease progression or relapse.
Disease control rate(DCR) | Up to 18 months from randomization date
  DCR is defined as the percentage of subjects who were evaluated for complete response(CR), partial response(PR), and stable disease(SD) as the best response among from randomization.
Quality of life(QoL) | after randomization(C1D1), D1 of every 3rd cycle(each cycle consists of 28 days) up to 18 months
  Evaluate changes compared to baseline using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
PK | The 12 eligible subjects will receive DHP107 and be taken blood samples for PK analysis on Day 1, 8 of Cycle 1
  Pharmacokinetics is defined as the study of the time course of drug absorption, distribution, metabolism, and excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Hope Rugo, M.D., Principal Investigator — University of California, San Francisco; David Weng, M.D., Principal Investigator — Anne Arundel Health System Research Institute (AAHS); Neelima Vidula, M.D., Principal Investigator — Massachusetts General Hospital (MGH); Adam Brufsky, M.D., Principal Investigator — University of Pittsburgh Medical Center (UPMC); Timothy Pluard, M.D., Principal Investigator — Saint Luke's Cancer Institute(SLCI); Priyanka Sharma, M.D., Principal Investigator — University of Kansas Medical Center(KUMC); Jane Skelton, M.D., Principal Investigator — Boca Raton Regional Hospital (BRRH); Richard Caradonna, M.D., Principal Investigator — ASCLEPES Research Center(ARC); Yan Ji, M.D., Principal Investigator — Metro-Minnesota Community Oncology Research Consortium (MMCORC); Craig Gordon, D.O., Principal Investigator — Michigan Center of Medical Research(MCMR); Ghassan Aljazayrly, M.D., Principal Investigator — California Research Institute (CRI); John Ellerton, M.D., Principal Investigator — Nevada Cancer Research Foundation (NCRF); Bohuslav Melichar, M.D., Principal Investigator — Onkologicka klinika, Fakultni nemocnice Olomouc (OUH); Martin Smakal, M.D., Principal Investigator — Onkologicky stacionar, NH Hospital a.s., nemocnice Horovice (NHH); Martina Zimovjanova, M.D., Principal Investigator — Onkologicka klinika, Vseobecna fakultni nemocnice v Praze (VFN)
Locations (15):
- United States (12):
  - California Research Institute (CRI), Los Angeles, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Boca Raton Regional Hospital (BRRH), Boca Raton, Florida
  - ASCLEPES Research Center(ARC), Weeki Wachee, Florida
  - Saint Luke's Cancer Institute(SLCI), Kansas City, Kansas
  - University of Kansas Medical Center(KUMC), Kansas City, Kansas
  - Anne Arundel Health System Research Institute (AAHS), Annapolis, Maryland
  - Massachusetts General Hospital(MGH), Boston, Massachusetts
  - Michigan Center of Medical Research(MCMR), Farmington Hills, Michigan
  - Metro-Minnesota Community Oncology Research Consortium (MMCORC), Minneapolis, Minnesota
  - Nevada Cancer Research Foundation (NCRF), Las Vegas, Nevada
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
- Czechia (3):
  - Onkologicka klinika, Fakultni nemocnice Olomouc (OUH), Olomouc, I.P. Pavlova 6
  - Onkologicky stacionar, NH Hospital a.s., nemocnice Horovice (NHH), Hořovice, K Nemocnici
  - Onkologicka klinika, Vseobecna fakultni nemocnice v Praze (VFN), Prague, U Nemocnice 499/2